CLINICAL TRIAL: NCT04740840
Title: Comparison of Anti-inflammatory Effects of Amlodipine and Levamlodipine in Patients With Hypertension
Brief Title: Anti Inflammatory Treatment of Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHNorthSichuanMC
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: Levamlodipine; Amlodipine; Serum inflammatory factors; Anti inflammatory treatment
MeSH Terms: conditions — Hypertension | interventions — levamlodipine; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levamlodipine group (Experimental): Blood pressure lowering therapy with 2.5mg levamlodipine, plus metoprolol succinate
  Interventions: Drug: Levamlodipine
- Amlodipine group (Sham Comparator): To receive 5mg amlodipine to lower blood pressure, plus metoprolol succinate
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Levamlodipine — According to the inclusion criteria of the trial, those who met the diagnosis of hypertension were randomly divided into the experimental group and the control group. The experimental group was treated with 2.5mg levamlodipine to lower blood pressure. Abdominal blood was emptying before the start of the trial and at the first and third month of medication.Data on CRP, TNF-α, IL-6, Lp-PLA2 and ATP were collected.
  Arms: Levamlodipine group
Drug: Amlodipine — According to the inclusion criteria, patients who met the diagnosis of hypertension were randomly divided into the experimental group and the control group. The experimental group was given 5mg amlodipine to lower blood pressure. Fasting blood was collected before the trial and during the first and third months of treatment. CRP, TNF-α, IL-6, Lp-PLA2 and ATP data were collected.
  Arms: Amlodipine group

SUMMARY:
To investigate the anti-inflammatory effect of amlodipine and levamlodipine in the treatment of hypertension

DETAILED DESCRIPTION:
A total of 200 inpatients or outpatients in the Department of cardiovascular medicine of the third people's Hospital of Mianyang City from April 2021 to October 2021, who met the diagnostic criteria of ish2020 international hypertension practice guidelines, were selected and randomly divided into control group and experimental group, with 100 cases in each group. The control group was treated with amlodipine and the experimental group was treated with levoamlodipine. The changes of blood pressure and serum inflammatory factors were observed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* ① In line with the diagnostic criteria of ISH2020 International Guidelines for Practice of Hypertension ② Age >18 years old, gender is not limited, during the treatment did not take other drugs that will affect blood pressure: such as antidepressants, oral contraceptives, Chinese herbal medicine, etc.; Voluntary participation and signing of informed consent, and can complete all the visit plan.

Exclusion Criteria:

* (1) Those who do not want to take blood tests; (2) Left ventricular ejection fraction < 50%, heart rate <50 beats/min; ③ Acute coronary syndrome (unstable angina pectoris and myocardial infarction); ④ valvular heart disease, congenital heart disease, etc.; Other infectious diseases and malignant tumors; ⑥ Bronchial asthma; ⑦ Abnormal liver function and renal dysfunction (ALT BBB 0 80U/L, CR BBB 1 442mmol/L); Autoimmune diseases or any serious and fatal diseases; ⑨ Receiving lipid-lowering therapy and oral vitamins or antioxidants; They are mentally ill, have no self-awareness, and are unable to express themselves or cooperate with others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2012-04-02 (Actual); Study Completion 2015-05-02 (Actual)

PRIMARY OUTCOMES:
After treatment, the blood pressure control of L-amlodipine group was better than that of amlodipine group | One month after treatment
the serum inflammatory factor level of L-amlodipine group was lower than that of amlodipine group | One month after treatment
Serum ATP level can be used to evaluate the anti-inflammatory effect of hypertension drugs | One month after treatment

IPD SHARING:
Plan to Share IPD: No